CLINICAL TRIAL: NCT05701657
Title: Nutrition for Precision Health, Powered by the All of Us Research Program
Brief Title: Nutrition for Precision Health, Powered by the All of Us
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of North Carolina, Chapel Hill (Other); Northwestern University (Other); Illinois Institute of Technology (Other); University of Chicago (Other); Pennington Biomedical Research Center (Other); Louisiana State University Health Sciences Center in New Orleans (Other); University of California, Davis (Other); University of California, Los Angeles (Other); Cedars-Sinai Medical Center (Other); University of Alabama at Birmingham (Other); Tufts University (Other); Massachusetts General Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); National Cancer Institute (NCI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); City University of New York, School of Public Health (Other); Mayo Clinic (Other); University of California, San Diego (Other); University of Hawaii (Other); Vanderbilt University Medical Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute of Drug Abuse (U.S. Federal Agency); Public Health Informatics Computational and Operations Research (Unknown); University of Southern California (Other); Cornell University (Other); University of Alabama, Tuscaloosa (Other); North Carolina State University (Other); University of North Carolina, Charlotte (Other); Duke University (Other); Stevens Institute of Technology (Other); Purdue University (Other); United States Military Academy West Point (U.S. Federal Agency); USDA, Western Human Nutrition Research Center (U.S. Federal Agency); North Carolina Central University (Other); Wake Forest University Health Sciences (Other); Boston University (Other); Children's Hospital of Richmond (Unknown); Virginia Commonwealth University (Other); Verily Life Sciences LLC (Industry); Indiana University (Other); Fred Hutchinson Cancer Center (Other); Columbia University (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00062970; UG1HD107692 (NIH); U24HD107676 (NIH); UG1HD107691 (NIH); UG1HD107697 (NIH); UG1HD107688 (NIH); UG1HD107696 (NIH); UG1HD107711 (NIH); U54TR004279 (NIH); U24CA268153 (NIH); U24DK131617 (NIH); U24CA268228 (NIH); U24OD023121 (NIH); OT2OD035404 (NIH); OT2OD030043 (NIH); AOD22022001 (Other Grant/Funding Number: National Institutes of Health (NIH) Inter Agency Agreement)
Record Dates: First submitted 2023-01-11; First posted 2023-01-27 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Nutrition; Health; Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Participants receive three standardized diets in a community-dwelling (Module 2) or live-in/residential settings (Module 3) setting.
Who Masked: Participant
Masking Description: Participants are masked to the 3 different diets (i.e., Diet A, Diet B, Diet C).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-Dwelling Controlled-Feeding Arm (Module 2) (Experimental): Participants drawn from Module 1 will receive three standardized diets (A, B, and C) in one of six sequences. Diet sequences are assigned at the cohort level based on a pre-defined site-specific schedule. All meals are provided while participants remain living in their own homes. Each diet period lasts ~14 days, separated by washouts of at least 14 days. Participants are masked to the nutritional content of each diet. Data collection includes wearable device outputs, physical and contextual assessments, and biospecimens. This arm evaluates metabolic responses to controlled diets under real-world, community-dwelling conditions.
  Interventions: Other: Diet A; Other: Diet B; Other: Diet C
- Residential Controlled-Feeding Arm (Module 3) (Experimental): A separate group of participants drawn from Module 1, who are not enrolled in Module 2, will receive the same three standardized diets administered in Module 2 while residing in a fully supervised residential setting. Diet sequences are assigned at the cohort level based on a pre-defined site-specific schedule. Each diet period will last approximately 14 days and will be separated by washout periods of at least 14 days. Intake, activity, and sleep will be closely monitored. Participants will also complete the same liquid meal test administered in Module 1 (see detailed description) after each of the diet periods. A wealth of measurements will be collected, including data from wearables, physical and contextual measures, and biospecimens. Intake balance studies are conducted in this module using the doubly labeled water assessments and DXA for body composition. Module 3 is designed to isolate the response to different diets from behavioral variability observed in community settings.
  Interventions: Other: Diet A; Other: Diet B; Other: Diet C

INTERVENTIONS:
Other: Diet A — This diet has high amounts of fruits/vegetables, whole grains, and beans, moderate amounts of dairy, meat/poultry/eggs, nuts/seeds, and olive oil, and very low amounts of sugar sweetened drinks and desserts.
Other: Diet B — This diet has high amounts of refined grains, meat/poultry/egg, sugar sweetened drinks, snacks, desserts, and processed foods. It has a moderate amount of dairy and low amounts of fruits/vegetables, whole grains, and fish.
Other: Diet C — This diet has moderate-high amounts of vegetables, meat/poultry/egg, nuts/seeds, dairy and fats/oils, low amounts of fruits, and very low amounts of grains and sugars.

SUMMARY:
The goal of this Nutrition for Precision Health (NPH) powered by All of Us research study is to develop Artificial Intelligence/Machine Learning (AI/ML) algorithms that predict individual responses to diet patterns using rich multimodal data streams collected across multiple domains (e.g., behavior, social, environmental, clinical and molecular biomarkers). NPH includes a large phenotyping cohort (Module 1, N=8000) and two separate follow-up groups drawn from a subset of Module 1participants. One group (Module 2, N=1200) receives three distinct diets in a 14-day crossover sequence, with at least a 14-day washout period between diets, while living in their own homes. A second group (Module 3, N=150) receives the same three diets under full-time supervision in a residential research setting. We will train and test AI/ML models to predict 0-4 hour postprandial response curves for glucose, insulin, triglycerides, and GLP-1, to the standardized diet-specific meal test (DSMT) collected after each of the three different diets delivered in Module 2. Each diet functions as a controlled stimulus to reveal biological features (such as individual variables, patterns, or clusters of measurements) that best predict a person's response.

The Module 2 DSMT response curves are the primary outcomes (dependent variables) for AI/ML algorithms that predict individual responses to diet patterns.

As a secondary objective, NPH will evaluate the validity and acceptability of technology-based dietary assessment tools. The Automated Self-Administered 24-hour recall (ASA24), Automatic Ingestion Monitor-2 (AIM-2), and the mobile food record (mFR) will be evaluated in Modules 2 and 3, and the ASA24 food record and the image-assisted ASA24 recall will be evaluated only in Module 3. Total energy intake, macronutrient and dietary fiber intake data are the main outcomes for validity testing compared against measures of actual intake. Acceptability will be determined from feedback surveys.

DETAILED DESCRIPTION:
The Nutrition for Precision Health (NPH) study is a multi-module, large-scale project with observational and interventional components embedded in the All of Us Research Program. The overarching goal is to develop artificial intelligence and machine learning (AI/ML) algorithms that predict individual responses to different diet patterns. The study consists of three modules designed to balance breadth (large scale phenotyping) and depth (controlled dietary interventions):

Module 1: Phenotyping (non-interventional)

Module 2: Community-dwelling controlled feeding group (Intervention arm 1)

Module 3: Residential (Live-in) controlled feeding group (Intervention arm 2)

Approximately 8,000 participants are anticipated to be enrolled in Module 1. From this cohort, approximately 1,200 participants will enroll in Module 2, and a separate subset of Module 1 participants (approximately 150 participants) will enroll in Module 3. Module 1 is observational and only Modules 2 and 3 are interventional in nature (intervention arms).

Module 1 is a phenotyping observational study. Participants undergo comprehensive characterization across an 8 to 10-day baseline period for assessments including: clinical measures, biospecimen collection, wearable sensor monitoring, questionnaires, and a liquid meal test (LMT). During the LMT, participants ingest a standardized liquid meal with a dose of acetaminophen for estimating gastric emptying and provide timed blood samples for postprandial profiling. The LMT is a diagnostic stimulus used solely for feature generation and is not being evaluated as an intervention. The resulting Module 1 high dimensional dataset supports machine learning methods (e.g., PCA, clustering, recursive feature elimination) for candidate predictor discovery and is therefore not listed in the Arms/Interventions section. Module 1 data will be used to develop novel statistical and machine learning methods to learn individual and generalizable causal models of nutrition and health, particularly in the presence of missing or incomplete data. The scale of Module 1 enables discovery of causal pathways and moderators between physical and contextual measures, LMT responses, and continuous glucose monitoring (CGM) data. These insights are critical for developing models that not only predict individual dietary responses but also explain why and under what conditions they occur.

Module 2 is a community dwelling controlled feeding arm (Intervention arm 1). A subset of Module 1 participants will enroll in Module 2, in which participants consume three standardized eucaloric diets; Diet A, Diet B, Diet C, in a crossover sequence. Each diet period lasts 12-14 days, separated by a minimum of 14-day washout period between diets. All meals are provided, but participants remain in their community dwelling environments. Participants undergo one of six possible sequences of dietary interventions, reflecting all possible orderings of the three diets (ABC, ACB, BCA, BAC, CAB, and CBA). To reduce potential bias, all six diet sequences are included in the crossover design. Rather than assigning diet sequences to individual participants, a cohort-based randomization approach is used to reduce operational burden on the metabolic kitchens. In this approach, pre-generated schedules involving all 6 diet sequences are randomly assigned to the clinical site metabolic kitchens, with each diet sequence corresponding to a cohort. Participants are then enrolled into the cohorts. The six diet orders are repeated over time at each site until the full enrollment targets for Modules 2 and 3 are met. Each site follows a different randomized version of the overall cohort schedule, which ensures distribution of the possible diet orders across time and clinical sites while preserving balance and logistical feasibility. Wearable-generated data (like accelerometry and CGM), physical and contextual measures are collected throughout.

At the completion of each diet participants are provided a standardized breakfast meal test, DSMT, from each of the three provided diets (Diet A, B, C). The 0-4 hour postprandial response curves are then used to evaluate inter-individual variation and unmask features collected in Module 1 and 2 that contribute to the AI/ML predictions of the response.

Each breakfast serves as a controlled stimulus to reveal underlying biological features from rich multimodal data streams, including clinical, molecular, behavioral, environmental, and social domains that may drive interindividual variability in metabolic response. For each DSMT, participants provide blood samples for up to nine time points over four hours. Analyte concentrations of glucose, insulin, triglycerides, and GLP-1, are used to construct response curves. The primary outcomes are the area under the curve (AUC) for each analyte (glucose, insulin, triglycerides, GLP-1) following each DSMT. This approach parallels a cardiac stress test: the stimulus (the meal) is a probe to expose individual variability in physiological function. Module 2 data will also be used to develop novel statistical and machine learning methods that produce individual and generalizable causal models of nutrition and health.

Module 3 is a controlled feeding study (Intervention arm 2) that is implemented in the live-in/residential setting. A separate subset of Module 1 participants completes the same three diets (Diet A, B, C) as in Module 2, but while residing in a research setting with full supervision of intake, activity, and sleep. The same cohort randomization scheme as in Module 2 determines diet order. The residential environment in Module 3 provides the highest degree of experimental control, allowing isolation of physiological effects of diet composition. Participants undergo a diet-specific meal test (DSMT) as well as a liquid meal test (LMT) accompanied by a dose of acetaminophen after completing each of the diets. In addition, intake balance studies are conducted in this module using the doubly labeled water assessments and DXA for body composition. Data from Module 3 will help quantify and separate variance in the AI/ML models attributable to adherence and other community dwelling factors observed in Module 2 and enables rigorous and controlled comparison against causal relationships discovered in Module 2 data.

In both Modules 2 and 3, participants are masked to the nutritional profile of each diet to minimize expectancy bias. Investigators and diet implementation staff are unmasked.

ELIGIBILITY:
Inclusion Criteria:

* Overall Inclusion -- Participants 18 years of age or older who have completed the primary All of Us consent process, Electronic Health Record consent process, have provided at least one All of Us biospecimen suitable for DNA sequencing, and have completed All of Us Participant Provided Information (PPI) Modules 1-3 (Basics, Overall Health, and Lifestyle); Speak English or Spanish; Able and willing to comply with study requirements and consent to participate.
* Module 1 -- Must be willing and able to comply with Module 1 protocol; Must provide informed consent for Module 1.
* Module 2 -- Must have completed Module 1; Must provide informed consent for Module 2; Must agree to comply with protocol over a period of approximately 10 to 12 weeks and up to six months. This includes consuming only the foods provided during periods of controlled feeding. Module 2 has three controlled feeding periods each lasting approximately two weeks with at least two weeks between feeding periods, and up to 6 months allowed for completion of the Module.
* Module 3 -- Must have completed Module 1; Must provide informed consent for Module 3; Must agree to comply with protocol over a period of approximately 10 to 12 weeks and up to 6 months. This includes being domiciled three times, for two weeks each, and consuming only the foods provided during the domiciled periods. There is at least two weeks between domiciled periods, and up to 6 months allowed for completion of the Module.

Exclusion Criteria:

* Module 1

  1. Any change to the participant's status from the time of All of Us enrollment that would render them ineligible for All of Us (e.g., being incarcerated, no longer living in the United States, or withdrawn from that study).
  2. Inability to provide informed consent and engage in informed consent procedures
  3. Participants who suffer from allergic reactions to, or are unwilling to consume, any components of the liquid mixed meal (e.g., milk products, soy products)
  4. Barriers to safe insertion of peripheral IV canula:

     1. Contraindications to peripheral IV canula insertion such as local skin infection, inflammation, trauma or burns if all the upper extremities were involved and there is no unaffected extremity available for IV placement; or
     2. A need for long-term IV access (e.g., ESRD); or
     3. Lymphedema or deep vein thrombosis (DVT) in the extremity of the IV (in the case where another extremity is not available); or
     4. Coagulopathy requiring blood thinning products; or
     5. Arteriovenous (AV) graft or fistula in the extremity of the IV (in the case where another extremity is not available)
  5. Pregnancy-related conditions:

     1. Gestational age precluding completion of the Module by 36 weeks. A pregnant participant should complete visit 1 by gestational age 34 weeks, 0 days and complete Module 1 by week 36.
     2. Severe morning sickness limiting mixed meal tolerance test (MMTT) consumption
  6. Certain types of disease states:

     1. Dumping syndrome or inability to consume the volume of the MMTT liquid
     2. Severe malabsorption such as history of short gut syndrome or need for parenteral or enteral nutrition
     3. Less than 12-months post-metabolic or bariatric surgery
     4. History of chronic pancreatitis (e.g., Cystic fibrosis) complicated by inability to tolerate the volume of the MMTT liquid
     5. Health conditions requiring chronic blood transfusions or iron infusions
     6. Hemoglobin <9.5 g/dL at screening
  7. Serious illness and in hospice or palliative care for terminal disease
  8. Swallowing issues:

     1. Self-reported difficulty tolerating solids or liquids
     2. Aspiration risks that require change in thickness of liquid or dietary modifications
  9. Short term antibiotic use. For example, active antibiotics use for an ongoing acute infection
  10. Blood donation in the last 3 months
  11. GLP-1 agonist medication (e.g. Semaglutide) instability as defined by less than 3 months of continuous use
  12. Any disorder, unwillingness, or inability not covered by any other exclusion criteria which, in the investigator's and/or team's opinion jeopardizes the safety of the participant or others or would interfere with adherence to the protocol.
* Module 2

  1. Any change to the participant's status from the time of All of Us enrollment that would render them ineligible for All of Us (e.g., being incarcerated, no longer living in the United States, or withdrawn from that study)
  2. All the above mentioned exclusion criteria for Module 1 (except inability to consume components of the liquid mixed meal)
  3. Inability to provide informed consent and engage in informed consent procedures
  4. Inability or failure to complete all critical elements from Module 1 (dietary, physical activity and sleep assessments, continuous glucose monitoring, MMTT)
  5. Participants who are already enrolled in Module 3
  6. Participants who are unlikely to be able to adhere to the protocol, based on structured adherence assessment by a study registered dietitian or other trained staff. This includes participants who have known allergic reactions to, or unwillingness to consume, study foods in Module 2 (e.g., gluten, meat, fish, nuts, dairy products) that cannot be reasonably accommodated by the metabolic kitchen within allowable criteria for the test diets.
  7. Participants who plan to relocate to an area not served by NPH or travel plans that do not permit completion of the Module over a period of up to 6 months.
  8. Pregnancy-related conditions:

     1. Gestational age precluding completion of the Module by week 36. A pregnant participant must be able to begin the first diet by gestational age 26 weeks, 0 days and complete the Module by week 36.
     2. High risk pregnancy defined as fetal anomaly, gestational hypertension (SBP >140 mmHg and DBP >90 mmHg), pre-eclampsia, or gestational diabetes mellitus
  9. Possible ethanol (alcohol) use disorder defined by Alcohol Use Disorders Identification Test (AUDIT) score of >15
  10. History of surgery for the treatment of obesity and:

      1. Self-reported dumping syndrome; or
      2. Following a special diet prescribed by their practitioner
  11. Uncontrolled disease states:

      1. Hypertension >160/100mmHg
      2. Exacerbation of underlying gastrointestinal disease, including inflammatory bowel disease or other malabsorptive disorders
      3. Decompensated cirrhosis
      4. Previously diagnosed diabetes Mellitus with HbA1c >12% at screening
      5. Newly diagnosed diabetes within the past three months, or HbA1c >6.5% at screening in a person not previously diagnosed with diabetes.
  12. Participants with a history of end-stage renal disease (ESRD) on hemodialysis
  13. Active infectious diseases (e.g., active tuberculosis < 3 months from symptom onset or positive test, COVID < 1 month from symptom onset or positive test)
  14. Malignancy (e.g., cancer) actively receiving cytotoxic chemotherapy (oral or infusions) treatment except for nonmelanoma skin cancers during the study period
  15. Participants who require dietary restrictions due to a medical condition or are on a prescribed diet for underlying chronic diseases
  16. Participants with type 1 or type 2 diabetes on insulin
  17. Participants aged ≥ 75 years with type 2 diabetes taking prescribed medications that can cause hypoglycemia (e.g. sulfonylureas, glinides), or on a prescribed diet
  18. Hospitalization for a chronic disease (e.g., congestive heart failure, stroke) within the past three months
  19. Requiring transfusions/apheresis during study period
  20. Participants with a current diagnosis of, or who have received treatment for, bulimia or anorexia nervosa within the past 3 years
  21. Participants with major psychiatric disorders, including major depression, schizophrenia, or psychosis, who have been hospitalized in the past six (6) months or are currently enrolled in treatment programs
  22. Hemoglobin <9.5 g/dL at screening
  23. Myocardial infarction, invasive cardiac procedure, participation in a cardiac or acute rehabilitation programs, transient ischemic attacks, or unstable arrhythmias within the past 3 months
  24. Any disorder, unwillingness, or inability not covered by any other exclusion criteria which, in the investigator's opinion, might jeopardize the safety of the participant or others, or be expected to interfere with adherence to the protocol.
* Module 3

  1. All the above mentioned exclusion criteria for Modules 1 and 2
  2. Participants who are already enrolled in Module 2
  3. Any disorder, unwillingness, or inability not covered by any other exclusion criteria which, in the investigator's opinion, might jeopardize the safety of the participant or others, or would interfere with adherence to the protocol
  4. Inability to abstain from tobacco or nicotine use, vaping, alcohol, illicit drug use, or recreational drug use for two (2) consecutive weeks while domiciled in the clinical unit. Nicotine gum, pouch, or patch are permitted.
  5. Any condition requiring in-person treatments or visits during the study period. This will not be accommodated by the domiciling protocol; however, tele-health visits with the participants regular doctor are permitted.
  6. Lactation or other infant care needs that cannot be accommodated while domiciled in the clinical unit
  7. Depression as assessed by:

     1. Patient Health Questionnaire (PHQ-9) score ≥ 15; or
     2. Affirmative answer to PHQ-9 suicidality question: "Thoughts that you would be better off dead or of hurting yourself in some way"
  8. Unable to engage in daily self-care activities (e.g., bathing, transferring, toileting, feeding, dressing)
  9. Uncontrolled endocrine disorders (such as Cushing's disease, pituitary disorders, diabetes)
  10. Uncontrolled pain requiring frequent or daily treatment, or adjustment of medication requiring weekly or bi-weekly visits. Pain medications used on an as-needed basis (PRN), such as acetaminophen or NSAIDs, are not excluded.
  11. Chronic prescription medications that would pose logistical and safety issues for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8000 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Glucose - Diet Specific mixed meal tolerance test (MMTT) Diet A | 4 hours
  Area under the curve (AUC) for glucose measured during the diet-specific MMTT for Diet A.
Insulin - Diet Specific mixed meal tolerance test (MMTT) Diet A | 4 hours
  Area under the curve (AUC) for insulin measured during the diet-specific MMTT for Diet A.
Triglycerides - Diet Specific mixed meal tolerance test (MMTT) Diet A | 4 hours
  Area under the curve (AUC) for triglycerides measured during the diet-specific MMTT for Diet A.
GLP-1 - Diet Specific mixed meal tolerance test (MMTT) Diet A | 4 hours
  Area under the curve (AUC) for Glucagon-Like Peptide-1 (GLP-1) measured during the diet-specific MMTT for Diet A.
Glucose - Diet Specific mixed meal tolerance test (MMTT) Diet B | 4 hours
  Area under the curve (AUC) for glucose measured during the diet-specific MMTT for Diet B.
Insulin - Diet Specific mixed meal tolerance test (MMTT) Diet B | 4 hours
  Area under the curve (AUC) for insulin measured during the diet-specific MMTT for Diet B.
Triglycerides - Diet Specific mixed meal tolerance test (MMTT) Diet B | 4 hours
  Area under the curve (AUC) for triglycerides measured during the diet-specific MMTT for Diet B.
GLP-1 - Diet Specific mixed meal tolerance test (MMTT) Diet B | 4 hours
  Area under the curve (AUC) for Glucagon-Like Peptide-1 (GLP-1) measured during the diet-specific MMTT for Diet B.
Glucose - Diet Specific mixed meal tolerance test (MMTT) Diet C | 4 hours
  Area under the curve (AUC) for glucose measured during the diet-specific MMTT for Diet C.
Insulin - Diet Specific mixed meal tolerance test (MMTT) Diet C | 4 hours
  Area under the curve (AUC) for insulin measured during the diet-specific MMTT for Diet C.
Triglycerides - Diet Specific mixed meal tolerance test (MMTT) Diet C | 4 hours
  Area under the curve (AUC) for triglycerides measured during the diet-specific MMTT for Diet C.
GLP-1 - Diet Specific mixed meal tolerance test (MMTT) Diet C | 4 hours
  Area under the curve (AUC) for Glucagon-Like Peptide-1 (GLP-1) measured during the diet-specific MMTT for Diet C.

SECONDARY OUTCOMES:
Accuracy of energy intake estimates from tool (ASA24, mFR, AIM-2, ASA24 record, mFR+ASA24) compared to known intake from objective measures. | 14 days
  Agreement will be assessed between total daily energy intake in kilocalories reported via each dietary assessment tool and known intake from the intake-balance method using doubly labelled water and provided diets.
Accuracy of energy intake estimates from tool (ASA24, mFR, AIM-2, ASA24 record, mFR+ASA24) compared to measured intake from provided diets. | 14 days
  Agreement between energy reported via each dietary assessment tool and measured intake from provided diets, in grams per day.
Accuracy of carbohydrate intake estimates from tool (ASA24, mFR, AIM-2, ASA24 record, mFR+ASA24) compared to measured intake from provided diets. | 14 days
  Agreement between carbohydrate intake reported via dietary assessment tool and measured intake from provided diets, in grams per day.
Accuracy of protein intake estimates from tool (ASA24, mFR, AIM-2, ASA24 record, mFR+ASA24) compared to measured intake from provided diets. | 14 days
  Agreement between protein intake reported via each dietary assessment tool and measured intake from provided diets, in grams per day.
Accuracy of fat intake estimates from tool (ASA24, mFR, AIM-2, ASA24 record, mFR+ASA24) compared to measured intake from provided diets. | 14 days
  Agreement between fat intake reported via each dietary assessment tool and measured intake from provided diets, in grams per day.
Accuracy of dietary fiber intake estimates from tool (ASA24, mFR, AIM-2, ASA24 record, mFR+ASA24) compared to measured intake from provided diets. | 14 days
  Agreement between dietary fiber intake reported via each dietary assessment tool and measured intake from provided diets, in grams per day.
Acceptability scales for ASA24 and Diet A | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for ASA24 and Diet B | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for ASA24 and Diet C | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for mFR and Diet A | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for mFR and Diet B | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for mFR and Diet C | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for AIM-2 and Diet A | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for AIM-2 and Diet B | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for AIM-2 and Diet C | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for ASA24 Record and Diet A | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for ASA24 Record and Diet B | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for ASA24 Record and Diet C | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for mFR+ASA24 and Diet A | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for mFR+ASA24 and Diet B | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."
Acceptability scales for mFR+ASA24 and Diet C | 14 days
  Responses to questions on ease of use and tool preference. Principal outcomes will be "ease of use" and "willingness to use again."

CONTACTS AND LOCATIONS:
Overall Officials: Marie G Gantz, PhD, Principal Investigator — RTI International
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - USDA Western Human Nutrition Research Center, Davis, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Davis, Sacramento, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - Northwestern University, Chicago, Illinois
  - Illinois Institute of Technology, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Tufts University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill - Chapel Hill Clinic, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill - Kannapolis, Kannapolis, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
IPD and related data dictionaries will be available in the All of Us Researcher Workbench.
Supporting Information: Study Protocol
Time Frame: One year after study completion
Access Criteria: Per the policies of the All of Us Research Workbench
URL: https://researchallofus.org/data-tools/workbench/